CLINICAL TRIAL: NCT02849431
Title: Mindfulness Approach for Adults Experiencing Borderline Personality Disorder; Supporting the Management of Intense and Fluctuating Emotions, a Feasibility Study
Brief Title: Mindfulness for Intense Emotions: A Feasibility Trial
Acronym: MindIE
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Unforeseen feasibility issues arose that meant the study did not seem viable in the current form.
Sponsor: Canterbury Christ Church University (Other)
Collaborators: Sussex Partnership NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 16/EM/0100
Record Dates: First submitted 2016-07-11; First posted 2016-07-29 (Estimated); Last update posted 2016-08-25 (Estimated); Status verified 2016-07

CONDITIONS: Borderline Personality Disorder
Keywords: mindfulness
MeSH Terms: conditions — Borderline Personality Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Mindfulness-based intervention (Experimental)
  Interventions: Behavioral: Mindfulness-based intervention

INTERVENTIONS:
Behavioral: Mindfulness-based intervention — A version of mindfulness-based cognitive therapy that has been adapted for people with a diagnosis of borderline personality disorder. This comprises eight weekly session, each lasting ninety minutes.

SUMMARY:
This study explores the feasibility of a mindfulness-based intervention for people with a diagnosis of borderline personality disorder.

DETAILED DESCRIPTION:
This is an uncontrolled feasibility trial of an eight-week mindfulness-based intervention for people with a diagnosis of borderline personality disorder. A battery of measures will be administered at baseline, in a time window of six to zero weeks prior to the start of the intervention. Outcome measures will be repeated in the two weeks after the end of the eight-week intervention, along with a qualitative interview.

ELIGIBILITY:
Inclusion criteria:

* Are on the caseload of a United Kingdom National Health Service Assessment and Treatment Service in the recruitment area and have had contact with that service in the past three months
* Have received the diagnosis of Borderline Personality Disorder from a suitably qualified health care professional, and continue to meet criteria for this diagnosis according to the SCID-II (Structured Clinical Interview for DSM Disorders Version II) at their screening assessment
* Have sufficient English language speaking and comprehension abilities to access group discussions and hand-out materials
* Have not previously engaged in a mindfulness-based intervention. As in other similar trials, a minimum dose has been operationally defined as having undertaken 50% or more of a mindfulness-based intervention delivered face-to-face by a suitably qualified health care professional
* Are not currently receiving, nor have plans to receive any other form of psychological therapy during the course of the study

Exclusion criteria:

* Have psychosis
* Misuse alcohol or drug to a level that requiring detox
* Have a intellectual disability
* Present a high level of risk requiring inpatient management at the time of their screening assessment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-07; Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Participant retention in percent | At post-intervention (i.e. 8 weeks after the start of the intervention).
  The number of participants who remain in the study at the post-intervention time point divided by the number of participants who are recruited into the study at baseline, expressed as a percentage

SECONDARY OUTCOMES:
Change from baseline at post-intervention in the Difficulties in the Emotion Regulation Scale (DERS) | Post-intervention (i.e. 8 weeks after the start of the intervention)
Change from baseline at post-intervention in the Patient Health Questionnaire (PQH-9). | Post-intervention (i.e. 8 weeks after the start of the intervention)
Change from baseline at post-intervention in the Generalized Anxiety Disorder Scale (GAD-7) | Post-intervention (i.e. 8 weeks after the start of the intervention)
Change from baseline at post-intervention in the Five-Facet Mindfulness Questionnaire (FFMQ) | Post-intervention (i.e. 8 weeks after the start of the intervention)
United Kingdom National Health Service Friends and Family Test (FFT). | Post-intervention (i.e. 8 weeks after the start of the intervention)
Elliot et al.'s (2001) Change Interview. | Post-intervention (i.e. 8 weeks after the start of the intervention)
Recruitment rate | Baseline
  The number of participants recruited into the study at baseline divided by the time taken to recruit these participants, measured from the date at which recruitment opened.
Qualitative feedback from participants on intervention acceptability in response to questions 6 and 7 of Elliot et al.'s (2001) Change Interview | Post-intervention (i.e. 8 weeks after the start of the intervention)

CONTACTS AND LOCATIONS:
Overall Officials: Hannah Droscher, Principal Investigator — Canterbury Christ Church University; Clara Strauss, Study Director — Sussex Partnership NHS Foundation Trust; Helen Startup, Study Director — Sussex Partnership NHS Foundation Trust; Fergal Jones, Study Director — Canterbury Christ Church University
Locations (1):
- Sussex Partnership NHS Foundation Trust, Brighton, Sussex, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Elliot R. (2012). Qualitative Methods for Studying Psychotherapy Change Processes. In: Thompson, A, & Harper D. (Eds.), Qualitative research methods in mental health and psychotherapy: An introduction for students and practitioners (pp. 69-81). Chichester, UK: Wiley-Blackwells